CLINICAL TRIAL: NCT06991686
Title: Prognostic Value of Procalcitonin Vs Platelet/Total Leukocytic Count Ratio in 28 Days Outcome in Severe Septic Patients
Brief Title: Comparison Between the Progostic Value of the Procalcitonin and the Platelet/Total Leukocytic Count Ratio in Sepsis
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MS 598/2024
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: All Conditions Causing Sepsis; Pneumonia - Bacterial; Urinary Tract Infection Bacterial
Keywords: sepsis; procalcitonin; prognosis; platelet/total leukocytic count ratio; outcome; prognostic value; septic patients
MeSH Terms: conditions — Pneumonia, Bacterial; Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood samples — blood sample for CBC and procalcitonin
Diagnostic Test: blood sample — blood sample for procalcitonin and CBC

SUMMARY:
What is already known on this subject? AND What does this study add? Sepsis is a complicated condition caused by a malfunction of the host's immune response to infection, which results in an uncontrollable inflammatory response and immunosuppression.

Sepsis is seen as a global health problem with significant economic effects .As a result, identifying prognostic and diagnostic biomarkers is critical in order to avoid adverse outcomes and reduce mortality by initiating treatment before irreversible damage occurs. A delay of one hour in sepsis treatment is thought to be associated with a 7-10 percent increase in sepsis-related death . As a result, many efforts have been made to find a viable biomarker for screening sepsis patients who are at a high risk of death.

Procalciotnin and platelet/leukocytic count ratio have been studied before but there are few studies comparing them.

Multiple studies have elucidated the benefits associated with the precursor molecule of calcitonin, specifically PCT, as a biomarker for sepsis.

In recent years, there has been a growing body of research indicating that platelets (PLT) and total leukocytic count are significant contributors to the inflammatory process. Previous research suggests a possible association between platelet/total leukocytic count ratio and sepsis mortality.

In this study will compare between the prognostic value of procalcitonin and the platelet/total leukocytic count ratio in sepsis.

AIM/ OBJECTIVES The aim of this prospective cross-sectional study was to compare the PCT level and the platelet/total leukocytic count ratio for survival prediction in patients with Sepsis.

METHODOLOGY:

* Type of Study: Prospective cross-sectional Study
* Study Setting: This study was conducted at Ain Shams University intensive care units.
* Study Period: Six months after approval of ethical committee of Faculty of Medicine, Ain Shams University or end of recruited sample size.

Sample Size:

Assuming an AUC for procalcitonin of 0.977 and that of platelet/total leukocytic count ratio of 0.944, a sample of 100 patients would be enough to detect such difference with 0.11 allowable difference between the 2 AUC, at 0.05 alpha error and 0.80 power of the test .

Ethical considerations

* The approval of the Scientific Research Ethics Committee at the Faculty of Medicine, Ain Shams University was obtained before starting work on the study.
* All data were considered confidential and weren't used outside this study without patient approval.
* Informed written consent was taken from all patients after explaining the study procedure in details.

Data collected and period of the study:

Clinical data and laboratory indicators, including gender, age, vital signs, past medical history such as hypertension and diabetes, SOFA score, APACHE II score, PLT, and PCT, were recorded within 24 hours of admission. Sepsis patients were observed and followed up for 28 days. Patient survival and death was recorded.

CBC was done every other day and serum procalcitonin was done every 72 hours for 28 days and the results were analysed and compared in correlation with patient's survivability.

Data management and analysis All data will be analyzed statistically. All data will be included in the SPSS software version 21. The appropriate statistical method will be used for analysis. Descriptive statistics such as mean, standard deviation and percentages will be used. Comparison of categorical data will be done using Chi-square test and for continuous data; unpaired "t" test will be used.

DETAILED DESCRIPTION:
What is already known on this subject? AND What does this study add? Sepsis is a complicated condition caused by a malfunction of the host's immune response to infection, which results in an uncontrollable inflammatory response and immunosuppression.

Sepsis is seen as a global health problem with significant economic effects . As a result, identifying prognostic and diagnostic biomarkers is critical in order to avoid adverse outcomes and reduce mortality by initiating treatment before irreversible damage occurs. A delay of one hour in sepsis treatment is thought to be associated with a 7-10 percent increase in sepsis-related death . As a result, many efforts have been made to find a viable biomarker for screening sepsis patients who are at a high risk of death.

Procalciotnin and platelet/leukocytic count ratio have been studied before but there are few studies comparing them.

In this study will compare between the prognostic value of procalcitonin and the platelet/total leukocytic count ratio in sepsis.

1. INTRODUCTION/ REVIEW Sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection, characterized by hypotension, elevated lactate, or oliguria. It is a common disease in critically ill patients and a major cause of death in intensive care units (ICUs). Despite improved understanding and management of sepsis over the past few decades, the mortality rate remains high, ranging from 20% to 45%, and it is a prominent challenge facing modern medicine and a significant global disease burden.

   Sepsis presents with a diverse range of clinical manifestations, and there is a lack of specific indicators for diagnosis and prognosis evaluation, and the disease progresses rapidly. As the condition worsens, there can be dysfunction of cellular metabolic processes, resulting in sepsis, multiple organ dysfunction syndrome, poor patient outcomes, and even death. Therefore, finding laboratory indicators that can quickly assist in diagnosing sepsis is one of the urgent problems to be solved in critical care medicine.

   A number of physicians have conducted research on the importance of blood biomarkers, including C-reactive protein, procalcitonin (PCT), and lactate, in the early evaluation of sepsis and in predicting patient outcomes.

   Multiple studies have elucidated the benefits associated with the precursor molecule of calcitonin, specifically PCT, as a biomarker for sepsis.

   In recent years, there has been a growing body of research indicating that platelets (PLT) and total leukocytic count are significant contributors to the inflammatory process. Previous research suggests a possible association between platelet/total leukocytic count ratio and sepsis mortality.

   Among all the sepsis biomarkers studied, complete blood count (CBC) metrics, including the platelet to total leukocytic count ratio , could be valuable tools . Undoubtedly, CBC has many advantages: (i) it is inexpensive, (ii) it has a quick turn-around time (TAT), (iii) it is accessible in all health centers, (iv) it is simple to perform, (v) clinicians regularly request CBC as part of patient management, and (vi) it is the most commonly ordered laboratory test in all medical settings, from the ICU to the emergency department (ED) Under inflammatory conditions, platelets (PLTs) have a role in promoting coagulation factor activation and cell aggregation, which can lead to host response dysregulation. When sepsis occurs, the inflammatory response of bacteria and platelets, endotoxin-mediated platelet activation, and the effects of circulating immune complexes can all lead to platelet reduction.Platelet reduction is one of the most common complications in sepsis patients, and it is negatively correlated with the severity of sepsis and mortality rates.

   Procalcitonin (PCT) is a nonhormonal glycoprotein whose levels are positively correlated with the severity of bacterial infections. It has important clinical significance in predicting the prognosis of infectious diseases and is a marker of disease course and treatment success. A multicenter randomized controlled trial involving sepsis patients showed that using PCT to guide patient antibiotic use can significantly reduce infection-related adverse events, 28-day mortality, and hospitalization costs.
2. AIM/ OBJECTIVES The aim of this prospective cross-sectional study was to compare the PCT level and the platelet/total leukocytic count ratio for survival prediction in patients with Sepsis.
3. METHODOLOGY:

   Patients and Methods/ Subjects and Methods/ Material and Methods
   * Type of Study: Prospective cross-sectional Study
   * Study Setting: This study was conducted at Ain Shams University intensive care units.
   * Study Period: Six months after approval of ethical committee of Faculty of Medicine, Ain Shams University or end of recruited sample size.

   Sample Size:

   Assuming an AUC for procalcitonin of 0.977 and that of platelet/total leukocytic count ratio of 0.944, a sample of 100 patients would be enough to detect such difference with 0.11 allowable difference between the 2 AUC, at 0.05 alpha error and 0.80 power of the test.

   Ethical considerations

   o The approval of the Scientific Research Ethics Committee at the Faculty of Medicine, Ain Shams University was obtained before starting work on the study.

   o All data were considered confidential and weren't used outside this study without patient approval.

   o Informed written consent was taken from all patients after explaining the study procedure in details.

   Study Tools and procedure:

   All patients included in this study were subjected on admission to the followings:

   A. History:
   * Personal data: name, age and gender.
   * Present history of medical condition.
   * Past medical history including:

     * Heart disease.
     * Liver disease
     * Renal disease
     * Hypertension.
     * Diabetes mellitus.
     * Hematological disorder.
     * Oncological disorder.

   B. Clinical examination:

   o Complete physical examination was done with emphasis on:

   - Vital signs: (heart rate, mean pressure, respiratory rate, temperature)

   - Mental status according to Glasgow Coma Score (GCS)

   - Chest examination.

   - Cardiac examination.

   - Abdominal examination.

   B. Clinical risk stratification:

   - APACHE II score SOFA score

   C. Laboratory investigations:

   Were done on admission and daily during the period of the study and included:

   - Serum Na, K.

   - Urea, creatinine.

   - Random blood sugar.

   - C-reactive protein.

   - Complete blood picture (Hemoglobin, White blood count (TLC), Platelet count).
   * Procalcitonin.

   D. Radiological examination that helps to detect source of sepsis included:
   * Chest X-ray.
   * Ultrasound of the abdomen.
   * CT abdomen with contrast.
   * Echo.

   E. Sepsis workup:
   * Blood cultures from one central and two peripheral lines.
   * Sputum culture or mini bronchio-alveolar lavage.
   * Urine culture.
   * Culture from a known source like abscess or tissue.

   F. Management:

   Management of all sepsis patients will be done according to the latest survival sepsis campaign guidelines including fluid resuscitation, vasopressor support and antimicrobial therapy.

   G. Data collected and period of the study:

   Clinical data and laboratory indicators, including gender, age, vital signs, past medical history such as hypertension and diabetes, SOFA score, APACHE II score, PLT, and PCT, were recorded within 24 hours of admission. Sepsis patients were observed and followed up for 28 days. Patient survival and death was recorded.

   CBC was done every other day and serum procalcitonin was done every 72 hours for 28 days and the results were analysed and compared in correlation with patient's survivability.

   Data management and analysis All data will be analyzed statistically. All data will be included in the SPSS software version 21. The appropriate statistical method will be used for analysis. Descriptive statistics such as mean, standard deviation and percentages will be used. Comparison of categorical data will be done using Chi-square test and for continuous data; unpaired "t" test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 21 years.
* Patients presented with sepsis defined as a suspected source of infection plus ≥2 of the following:

  * Fever of >38º or hypothermia <36º
  * Heart rate of >90 beats/min
  * Respiratory rate of >20 breaths per minute or PaCO2 <32 mmHg
  * White blood cells >12 x 109/cmm or <4 x 109/cmm, or >10% immature forms.
* Patients presented with severe sepsis defined as sepsis associated with secondary organ dysfunction.

Exclusion Criteria:

* Age less than 21 years.
* Patients with acute cerebro-vascular event.
* Patients on chemotherapy.
* Patients with malignant hematological disease.
* Patients with immunosuppression.
* Patients with active hemorrhage.
* Patients who had used anti-PLT drugs such as clopidogrel prior to admission.
* Patients with life threating medical comorbidities (e.g.intractable heart failure, hepatic encephalopathy).
* Patients diagnosed with heparin induced thrombocytopenia (HIT).
* Patients on medications that help reducing platelet count such as linezolid.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was carried out on adult critically ill patients of both sexes with sepsis whom admitted to the Critical Care units of Ain Shams University Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
mortality | 28 days
  survival or death of the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Meidcine Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Shannon O. The role of platelets in sepsis. Res Pract Thromb Haemost. 2020 Dec 20;5(1):27-37. doi: 10.1002/rth2.12465. eCollection 2021 Jan. PMID 33537527
- [Background] Standage SW, Wong HR. Biomarkers for pediatric sepsis and septic shock. Expert Rev Anti Infect Ther. 2011 Jan;9(1):71-9. doi: 10.1586/eri.10.154. PMID 21171879
- [Background] Kim H, Kim Y, Lee HK, Kim KH, Yeo CD. Comparison of the delta neutrophil index with procalcitonin and C-reactive protein in sepsis. Clin Lab. 2014;60(12):2015-21. doi: 10.7754/clin.lab.2014.140528. PMID 25651736
- [Background] de Souza DC, Machado FR. Epidemiology of Pediatric Septic Shock. J Pediatr Intensive Care. 2019 Mar;8(1):3-10. doi: 10.1055/s-0038-1676634. Epub 2018 Dec 28. PMID 31073502
- [Background] Huang M, Cai S, Su J. The Pathogenesis of Sepsis and Potential Therapeutic Targets. Int J Mol Sci. 2019 Oct 29;20(21):5376. doi: 10.3390/ijms20215376. PMID 31671729
- [Background] Paoli CJ, Reynolds MA, Sinha M, Gitlin M, Crouser E. Epidemiology and Costs of Sepsis in the United States-An Analysis Based on Timing of Diagnosis and Severity Level. Crit Care Med. 2018 Dec;46(12):1889-1897. doi: 10.1097/CCM.0000000000003342. PMID 30048332
- [Background] Andersson P, Frigyesi A. High-sensitivity troponin T is an important independent predictor in addition to the Simplified Acute Physiology Score for short-term ICU mortality, particularly in patients with sepsis. J Crit Care. 2019 Oct;53:218-222. doi: 10.1016/j.jcrc.2019.06.018. Epub 2019 Jun 19. PMID 31277048
- [Background] Rello J, Valenzuela-Sanchez F, Ruiz-Rodriguez M, Moyano S. Sepsis: A Review of Advances in Management. Adv Ther. 2017 Nov;34(11):2393-2411. doi: 10.1007/s12325-017-0622-8. Epub 2017 Oct 11. PMID 29022217
- [Background] Agnello L, Giglio RV, Bivona G, Scazzone C, Gambino CM, Iacona A, Ciaccio AM, Lo Sasso B, Ciaccio M. The Value of a Complete Blood Count (CBC) for Sepsis Diagnosis and Prognosis. Diagnostics (Basel). 2021 Oct 12;11(10):1881. doi: 10.3390/diagnostics11101881. PMID 34679578